CLINICAL TRIAL: NCT00744939
Title: Prospective Non-randomized Observational (Pharmacoepidemiologic) Cohort Study (Open-label, Multicenter) to Assess the Magnitude of Potential Risk With the Administration of Magnevist® Injection in Patients With Moderate Renal Impairment for the Development of Nephrogenic Systemic Fibrosis (NSF) Based on Diagnostically Specific Clinical and Histopathologic Information.
Brief Title: Risk of Nephrogenic Systemic Fibrosis (NSF) in Patients With Moderate Renal Insufficiency After the Administration of Magnevist
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 13256; X312141 (Other: Company internal)
Record Dates: First submitted 2008-08-20; First posted 2008-09-01 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Fibrosis; Kidney Failure; Renal Insufficiency
Keywords: Gadolinium; NSF; Renal Impairment; chemically induced; adverse effects; Contrast Media; complications
MeSH Terms: conditions — Fibrosis; Renal Insufficiency | interventions — Gadolinium DTPA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum creatinine must be obtained within 6 weeks of the administration of Magnevist, or as currently recommended by the American College of Radiology. At the Baseline within 48 hrs. pre-injection a chemistry panel will be obtained in all patients after intravenous access has been obtained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Gadopentetate dimeglumine (Magnevist, BAY86-4882): Participants received Magnevist in accordance with its labeling
  Interventions: Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882)

INTERVENTIONS:
Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882) — Patients will be followed for 2 years after the administration of Magnevist at the approved dose to see if symptoms consistent with NSF develop

SUMMARY:
Assess potential risk for NSF in subjects with renal impairment (moderate) post magnevist injection. Subjects will be screened within 48 hours of previously scheduled MRI, those meeting the enrollment criteria will be enrolled prior to MRI and followed for 2 years post MRI with visits occuring at 1yr and 2 yr timepoints, in addition follow-up phone calls conducted at 1, 3, 6 and 18 months to assess for skin changes suggestive of NSF.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have moderate (eGFR 30-59 ml/min/1.73 m^2) renal impairment and be scheduled for a contrast enhanced MRI with Magnevist Injection at the recommended dose of 0.1 mmol/kg.

Exclusion Criteria:

* Gadolinium Based Contrast Agent (other then Magnevist) enhanced MRI within 12 months prior to administration of Magnevist
* History of NSF
* Clinically unstable or age <2 yrs

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who are scheduled to undergo CE-MRI with Magnevist and for which the inclusion and exclusion criteria are fulfilled are eligible for enrolment into the study.
Sampling Method: Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2008-11; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (22):
- United States (22):
  - Phoenix, Arizona
  - Chula Vista, California
  - Los Angeles, California
  - Santa Rosa, California
  - Pueblo, Colorado
  - New Haven, Connecticut
  - Jacksonville, Florida
  - Honolulu, Hawaii
  - Topeka, Kansas
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Brooklyn, New York
  - New York, New York
  - Stony Brook, New York
  - Cleveland, Ohio
  - Danville, Pennsylvania
  - Philadelphia, Pennsylvania
  - Memphis, Tennessee
  - Houston, Texas
  - San Antonio, Texas
  - Charlottesville, Virginia
  - Tacoma, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant's first visit was on 21 Nov 2008. Nineteen study centers in the United States screened and enrolled participants scheduled to undergo contrast enhanced magnetic resonance imaging (CE-MRI) with Magnevist within the approved indications at the recommended dose of 0.1 mmol/kg body weight.
Pre-assignment Details: A total of 168 participants were enrolled.
Period: Overall Study
Arm/Group | Gadopentetate Dimeglumine (Magnevist, BAY86-4882)
Started | 168
Treatment Received | 141
Completed | 77
Not Completed | 91
Not completed — Withdrawal by Subject | 9
Not completed — Protocol Violation | 13
Not completed — Death | 24
Not completed — distance | 4
Not completed — Lost to Follow-up | 12
Not completed — Medical history exclusionary | 1
Not completed — Did not receive Magnevist | 7
Not completed — Failed inclusion/exclusion criteria | 19
Not completed — coma | 1
Not completed — incorrect race | 1

BASELINE CHARACTERISTICS:
Groups:
- Mild Renal Impairment: Participants with estimated glomerular filtration rate (eGFR) >65 mL/min/1.73 m^2 prior to Magnevist injection was classified into cohort of Mild renal impairment.
- Extended Moderate Renal Impairment: Participants with eGFR between >59 and ≤65 mL/min/1.73 m^2 prior to Magnevist injection was classified into cohort of extended moderate renal impairment.
- Moderate Renal Impairment: Participants with eGFR between ≥30 and ≤59 mL/min/1.73 m^2 prior to Magnevist injection was classified into cohort of moderate renal impairment.
- Severe Renal Impairment: Participants on dialysis or subjects with eGFR <30 mL/min/1.73 m^2 prior to Magnevist injection was classified into cohort of severe renal impairment.
- Total: Total of all reporting groups
Arm/Group | Mild Renal Impairment | Extended Moderate Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment | Total
Number analyzed (Participants) | 14 | 9 | 109 | 9 | 141
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.0 (12.03) | 66.9 (9.91) | 66.4 (12.09) | 62.4 (9.51) | 66.0 (11.75)
Age, Customized [Number; unit: Participants]
  <65 years | 5 | 5 | 47 | 6 | 63
  >=65 years | 9 | 4 | 62 | 3 | 78
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 52 | 4 | 62
  Male | 11 | 6 | 57 | 5 | 79
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 7 | 0 | 9
  Not Hispanic or Latino | 13 | 8 | 102 | 9 | 132
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 5 | 0 | 5
  Black or African American | 2 | 0 | 18 | 1 | 21
  White | 11 | 9 | 81 | 8 | 109
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 3 | 0 | 3
Weight [Mean (Standard Deviation); unit: Kilograms] — Overall number of baseline participants for moderate cohort is 107
  Kilograms | 85.2 (13.1) | 81.9 (13.3) | 86.0 (18.3) | 83.2 (18.4) | 85.5 (17.5)
Years since renal diagnosis [Mean (Standard Deviation); unit: Years] — Number of participants with information available: mild cohort is 5;extended moderate cohort is 1; moderate cohort is 38 ; severe cohort 3.
  Years | 4.4 (4.5) | 0 (0) | 2.2 (3.2) | 3.1 (4.6) | 2.4 (3.4)
Cause of renal disease [Number; unit: Participants] — Participants might have more than one cause of renal disease reported.
  Participants
    Diabetes | 3 | 2 | 28 | 5 | 38
    Glomerulonephritis | 0 | 0 | 1 | 0 | 1
    Collagen disease | 0 | 0 | 0 | 0 | 0
    Hypertension | 7 | 3 | 41 | 2 | 53
    Polycystic kidney disease | 0 | 0 | 3 | 2 | 5
    Other | 8 | 5 | 68 | 3 | 84
Receiving dialysis [Number; unit: Participants] — Not all participants were receiving dialysis at baseline.
  Participants
    Any | 0 | 0 | 0 | 2 | 2
    Peritoneal dialysis | 0 | 0 | 0 | 0 | 0
    Hemodialysis | 0 | 0 | 0 | 2 | 2
Vascular injuries [Number; unit: Participants] — Participants reporting more than one injury per injury type were counted only once for each type. Not all patients had vascular injuries reported.
  Participants
    Any | 3 | 1 | 36 | 3 | 43
    Shunt surgery/repair | 0 | 0 | 4 | 2 | 6
    Organ transplant surgery | 0 | 0 | 5 | 3 | 8
    Thrombotic events | 1 | 1 | 24 | 0 | 26
    Other surgeries | 2 | 0 | 13 | 0 | 15
    Other | 0 | 0 | 4 | 0 | 4
MRI region of main interest [Number; unit: Participants]
  Brain | 4 | 3 | 28 | 1 | 36
  Spine | 1 | 0 | 11 | 1 | 13
  Liver | 1 | 1 | 19 | 3 | 24
  Kidney | 2 | 2 | 15 | 1 | 20
  Musculoskeletal | 1 | 0 | 8 | 0 | 9
  Other | 5 | 3 | 28 | 3 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed Nephrogenic Systemic Fibrosis (NSF), Based on Diagnostically Specific Clinical and Histopathological Information-cohort Analysis and Full Analysis Set
Description: Either clinical or histopathology score had to be at least 2 and the other at least 3 for diagnosis of NSF. Clinical score 2, 3 or 4 was derived from more than one minor criterion finding, one major criterion finding or more than one major criterion finding respectively. Major Criteria include patterned plaques, joint contractures, cobblestoning and marked induration/Peau d'orange (upper extremity or above knee); minor Criteria include puckering/linear banding, superficial (plaque/patch), dermal papules and scleral plaques (subject aged <45 years). Pathology score 2, 3 or 4 was derived from 2, 3 or at least 4 histological criteria findings respectively. Histological Criteria include increased cellularity (spindled and/or epithelioid) with few other inflammatory cells, CD34+ spindle or epithelioid cells in a reticular or parallel arrangement with "tram-tracking," presence of both fine collagen and ropey collagen surrounded by clefts, elastic fibers preserved and septal involvement.
Time Frame: Up to 24 months following the administration of Magnevist
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Mild Renal Impairment | Extended Moderate Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 14 | 9 | 109 | 9
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants Who Developed NSF, Based on Diagnostically Specific Clinical and Histopathological Information-full Analysis Set
Description: as for outcome 1
Time Frame: Up to 24 months following the administration of Magnevist
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine (Magnevist, BAY86-4882)
Number analyzed (Participants) | 141
Participants | 0

3. Primary Outcome: Number of Participants Who Developed NSF, Based on Diagnostically Specific Clinical and Histopathological Information-cohort Analysis and Per Protocol Set
Description: as for outcome 1
Time Frame: Up to 24 months following the administration of Magnevist
Population: Per Protocol Set. Participants with mild and extended moderate renal impairment were excluded from the per protocol analysis.
Measure: Number; unit: Participants
Arm/Group | Mild Renal Impairment | Extended Moderate Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 0 | 0 | 58 | 8
Participants |  |  | 0 | 0

4. Primary Outcome: Number of Participants Who Developed NSF, Based on Diagnostically Specific Clinical and Histopathological Information-per Protocol Set
Description: as for outcome 1
Time Frame: Up to 24 months following the administration of Magnevist
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine (Magnevist, BAY86-4882)
Number analyzed (Participants) | 66
Participants | 0

5. Secondary Outcome: Total Number of Participants With Clinicopathological Correlation of 'NSF' or 'Consistent With NSF' and Subjects Without Biopsy Developing Clinical Signs Consistent With NSF-cohort Analysis and Full Analysis Set
Description: Either clinical or histopathology score need at least 2 and the other at least 3 for diagnosis of NSF. Clinical score 2, 3 or 4 required more than 1 minor criterion, 1 major criterion or more than 1 major criterion respectively. Major criteria: patterned plaques, joint contractures, cobblestoning, marked induration/Peau d'orange (upper extremity or above knee); minor Criteria: puckering/linear banding, superficial (plaque/patch), dermal papules, scleral plaques (subject aged <45 yrs). Pathology score 2, 3 or 4 required 2, 3 or at least 4 histological criteria respectively. Histological criteria include Increased cellularity with few other inflammatory cells, CD34+ spindle or epithelioid cells in a reticular or parallel arrangement with "tram-tracking," presence of fine collagen and ropey collagen surrounded by clefts, elastic fibers preserved and Septal involvement. A clinical score of 4 was suggestive of developing clinical signs consistent with NSF in subjects without biopsy.
Time Frame: Up to 24 months following the administration of Magnevist
Population: Full analysis set
Measure: Number; unit: Participants
Groups:
- Extended Moderate Renal impairmentEdit: Subjects with eGFR between >59 and ≤65 mL/min/1.73 m2 prior to Magnevist injection was classified into cohort of extended moderate renal impairment
Arm/Group | Mild Renal Impairment | Extended Moderate Renal impairmentEdit | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 14 | 9 | 109 | 9
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Total Number of Participants With Clinicopathological Correlation of 'NSF' or 'Consistent With NSF' and Subjects Without Biopsy Developing Clinical Signs Consistent With NSF-full Analysis Set
Description: as for outcome 5
Time Frame: Up to 24 months following the administration of Magnevist
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine (Magnevist, BAY86-4882)
Number analyzed (Participants) | 141
Participants | 0

7. Secondary Outcome: Total Number of Participants With Clinicopathological Correlation of 'NSF' or 'Consistent With NSF' and Subjects Without Biopsy Developing Clinical Signs Consistent With NSF-cohort Analysis and Per Protocol Set
Description: as for outcome 5
Time Frame: Up to 24 months following the administration of Magnevist
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Mild Renal Impairment | Extended Moderate Renal impairmentEdit | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 0 | 0 | 58 | 8
Participants |  |  | 0 | 0

8. Secondary Outcome: Total Number of Participants With Clinicopathological Correlation of 'NSF' or 'Consistent With NSF' and Subjects Without Biopsy Developing Clinical Signs Consistent With NSF-per Protocol Set
Description: Either clinical or histopathology score need at least 2 and the other at least 3 for diagnosis of NSF. Clinical score 2, 3 or 4 required more than 1 minor criterion, 1 major criterion or more than 1 major criterion respectively. Major criteria: patterned plaques, joint contractures, cobblestoning, marked induration/Peau d'orange (upper extremity or above knee); minor Criteria: puckering/linear banding, superficial (plaque/patch), dermal papules, scleral plaques (subject aged <45 yrs). Pathology score 2, 3 or 4 required 2, 3 or at least 4 histological criteria respectively. Histological criteria include Increased cellularity with few other inflammatory cells, CD34+ spindle ore epithelioid cells in a reticular or parallel arrangement with "tram-tracking," presence of fine collagen and ropey collagen surrounded by clefts, elastic fibers preserved and Septal involvement. A clinical score of 4 was suggestive of developing clinical signs consistent with NSF in subjects without biopsy.
Time Frame: Up to 24 months following the administration of Magnevist
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine (Magnevist, BAY86-4882)
Number analyzed (Participants) | 66
Participants | 0

9. Secondary Outcome: Number of Participants With Adverse Events (AEs) Reported in Association With the Administration of Magnevist-cohort Analysis and Full Analysis Set
Description: Adverse events occurring within 1 day after administration of Magnevist or skin-related adverse events occurring during follow-up (FU) were recorded.
Time Frame: Up to 24 months following the administration of Magnevist
Population: Full analysis set.
Measure: Number; unit: Participants
Arm/Group | Mild Renal Impairment | Extended Moderate Renal impairmentEdit | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 14 | 9 | 109 | 9
Participants
  Participants with AEs within 1 day | 0 | 0 | 0 | 0
  Participants with skin-related AEs during FU | 0 | 3 | 12 | 0

10. Secondary Outcome: Number of Participants With Adverse Events (AEs) Reported in Association With the Administration of Magnevist-full Analysis Set
Description: as for outcome 9
Time Frame: Up to 24 months following the administration of Magnevist
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine (Magnevist, BAY86-4882)
Number analyzed (Participants) | 141
Participants
  Participants with AEs within 1 day | 0
  Participants with skin-related AEs during FU | 15

11. Secondary Outcome: Number of Participants With Adverse Events (AEs) Reported in Association With the Administration of Magnevist-cohort Analysis and Per Protocol Set
Description: as for outcome 9
Time Frame: Up to 24 months following the administration of Magnevist
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Mild Renal Impairment | Extended Moderate Renal impairmentEdit | Moderate Renal Impairment | Severe Renal Impairment
Number analyzed (Participants) | 0 | 0 | 58 | 8
Participants
  Participants with AEs within 1 day |  |  | 0 | 0
  Participants with skin related AEs during FU |  |  | 7 | 0

12. Secondary Outcome: Number of Participants With Adverse Events (AEs) Reported in Association With the Administration of Magnevist-per Protocol Set
Description: as for outcome 9
Time Frame: Up to 24 months following the administration of Magnevist
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Gadopentetate Dimeglumine (Magnevist, BAY86-4882)
Number analyzed (Participants) | 66
Participants
  Participants with AEs within 1 day | 0
  Participants with skin-related AEs during FU | 7

ADVERSE EVENTS:
Time Frame: Up to 24 months following the administration of Magnevist
Groups:
- Mild Renal Impairment: Participants with eGFR >65 mL/min/1.73 m^2 prior to Magnevist injection was classified into cohort of Mild renal impairment.
Arm/Group | Mild Renal Impairment | Extended Moderate Renal Impairment | Moderate Renal Impairment | Severe Renal Impairment
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/9 | 1/109 | 0/9
Other Adverse Events (participants affected / at risk) | 0/14 | 3/9 | 12/109 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Renal Impairment (N=14) | Extended Moderate Renal Impairment (N=9) | Moderate Renal Impairment (N=109) | Severe Renal Impairment (N=9)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mild Renal Impairment (N=14) | Extended Moderate Renal Impairment (N=9) | Moderate Renal Impairment (N=109) | Severe Renal Impairment (N=9)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Bayer HealthCare was informed about the release from the postmarketing surveillance (PMS) for Magnevist with a letter dated 02 JUN 2011. As a consequence Bayer HealthCare stopped enrollment for this study on 01 AUG 2011.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No